CLINICAL TRIAL: NCT04067453
Title: External Anal Sphincter Fatigability, an Electromyographic and Manometric Study
Brief Title: External Anal Sphincter Fatigability
Acronym: EASF
Status: Completed | Type: Observational
Sponsor: Gérard Amarenco (Other)
Responsible Party: Sponsor-Investigator, Gérard Amarenco, Head of Neuro-Urology department, Tenon Hospital, Pierre and Marie Curie University
Organization: Pierre and Marie Curie University (Other)
Other Study IDs: GRC--01 GREEN
Record Dates: First submitted 2019-08-12; First posted 2019-08-26 (Actual); Last update posted 2019-11-29 (Actual); Status verified 2019-11

CONDITIONS: External Anal Sphincter Fatigability
Keywords: Anal Canal; External Anal Sphincter; Muscle fatigue; Electromyography; Anorectal Manometry

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients undergoing fatiguing protocol: patient consulting for anorectal manometry in order to explore anorectal disorders with a voluntary command on external anal sphincter
  Interventions: Other: Fatiguing contractions

INTERVENTIONS:
Other: Fatiguing contractions — 10 sustained external anal sphincter contractions with maximal voluntary contraction of 20 seconds followed by 10 seconds of resting.

SUMMARY:
External anal sphincter is a Skeletal muscle under voluntary control. As described in previous studies, it is mainly composed of type 1 fibers. Fatigability is a concept which has been studied and described many times in skeletal limbs muscles. Two types of fatigue are described, peripheral of central fatigue. Fatigue can been physiologic but also pathologic (due to an affection of the muscle, the peripheral nervous system or the central nervous system). Many tools have been used to measure muscle fatigability (direct strength measure on isometric contraction, electromyography, echography, oxymetry...).

Besides many fatiguing methods have been developed for every each muscle depending on its histological structure.

Anal sphincter fatigability has already been described in few manometric studies with particularly 2 measures: Fatigue Rate and Fatigue Rate Index. Moreover, no fatiguing protocol has been standardized to study it.

The primary aim of this study is to define a fatiguing protocol for external anal sphincter in order to study it in further studies. Secondary aims are to assess Electromyography as a tool for measuring this fatigability and finally to assess the link between anal sphincter fatigability and symptoms reported by patients.

Patients over 18 years old, consulting for an Anorectal Manometry with a voluntary command on the external anal sphincter are included.

History and treatment, height, weight, sex, age, Fatigue impact scale, digestive symptoms with Neurologic Bowel Disorders score and Wexner scale, urinary tract symptoms with Urinary Symptom Profile (USP) score and electromyography (Root Mean Square (RMS) and Mean Power Frequency (MPF)) and manometric data (contraction peak, fatigue rate, fatigue rate index) were recorded.

The fatiguing protocol consists in 10 sustained external anal sphincter contractions with maximal voluntary contraction of 20 seconds followed by 10 seconds of resting. A training contraction is made before the fatiguing protocol. At the end of the protocol, patients undergo a classical anorectal manometry.

Primary outcome is the difference on root mean square in electromyography between the first and the last fatiguing contraction.

Secondary outcomes were mean power frequency and manometric data (i.e. Fatigue Rate index (FRI), Fatigue Rate (FR), contraction Peak)

Influence of age, sex, symptoms, pathologies, weight on fatigability will be studied in a second analysis

ELIGIBILITY:
Inclusion Criteria:

* over 18 years old
* voluntary command on external anal sphincter contraction during physical examination
* Anorectal disorders

Exclusion Criteria:

* inability to understand simple orders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all patients over 18 years old presenting for anorectal manometry examination in order to explore anorectal disorders between 01/08/2019 and 31/10/2019 with a voluntary command on external anal sphincter contraction
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2019-11-02 (Actual)

PRIMARY OUTCOMES:
Variation in electromyographic muscle response 1 | 1 day
  Difference between first and last fatiguing contractions on surface electromyographic Root Mean Square (RMS)

SECONDARY OUTCOMES:
variation of electromyographic muscle response 2 | 1 day
  Difference between first and last fatiguing contractions on surface electromyographic Mean Power Frequency (MPF)
variation of external anal sphincter contractions with manometry 1 | 1 day
  Difference between first and last contractions on manometrical Fatigue rate
variation of external anal sphincter contractions with manometry 2 | 1 day
  Difference between first and last contractions on manometrical Fatigue rate Index
variation of external anal sphincter contractions with manometry 3 | 1 day
  Difference between first and last contractions on manometrical Peak of Contraction

CONTACTS AND LOCATIONS:
Overall Officials: Gérard Amarenco, Principal Investigator — Study Principal Investigator Sorbonne Université, GRC 001, GREEN, AP-HP, Hôpital Tenon, Paris, France
Locations (1):
- department of Neuro-Urology, Hôpital Tenon, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided